CLINICAL TRIAL: NCT00947882
Title: A Dose-Finding, Multi-Centre, Double-Blind, Randomised, Parallel, Placebo-Controlled Trial to Investigate Efficacy and Safety of Degarelix in Men With Lower Urinary Tract Symptoms (LUTS) Associated With Benign Prostatic Hyperplasia (BPH)
Brief Title: A Trial of Degarelix in Men With Lower Urinary Tract Symptoms (LUTS) Associated With Benign Prostatic Hyperplasia (BPH)
Acronym: DELUTS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FE200486 CS36; 2009-012325-11 (EudraCT Number); 104367 (Other: IND Number)
Record Dates: First submitted 2009-07-27; First posted 2009-07-28 (Estimated); Results first posted 2015-05-14 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-05

CONDITIONS: Lower Urinary Tract Symptoms (LUTS)
MeSH Terms: conditions — Lower Urinary Tract Symptoms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Degarelix 10 mg (Experimental)
  Interventions: Drug: Degarelix 10 mg
- Degarelix 20 mg (Experimental)
  Interventions: Drug: Degarelix 20 mg
- Degarelix 30 mg (Experimental)
  Interventions: Drug: Degarelix 30 mg

INTERVENTIONS:
Drug: Placebo — Mannitol 50 mg/mL solution
  Arms: Placebo
Drug: Degarelix 10 mg — 10 mg degarelix, 40 mg/mL solution
  Other Names: FE200486; Firmagon
  Arms: Degarelix 10 mg
Drug: Degarelix 20 mg — 20 mg degarelix, 40 mg/mL solution
  Other Names: FE200486; Firmagon
  Arms: Degarelix 20 mg
Drug: Degarelix 30 mg — 30 mg degarelix, 40 mg/mL solution
  Other Names: FE200486; Firmagon
  Arms: Degarelix 30 mg

SUMMARY:
A dose-finding, multi-centre, double-blind, randomised, parallel, placebo-controlled trial to investigate efficacy and safety of degarelix in men with lower urinary tract symptoms (LUTS) associated with benign prostatic hyperplasia (BPH)

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained before any trial-related activity is performed
* Men, aged 50 or older
* Clinical signs and symptoms of BPH for ≥6 months
* Moderate to severe LUTS at screening, as defined by International Prostate Symptom Score (IPSS) ≥13
* An IPSS QoL score of ≥3 at screening
* Prostate specific antigen (PSA) at screening ≤10 ng/mL (responsibility of the Investigator to rule out prostate cancer when PSA is >4 ng/mL, except in the USA where patients with a PSA >4 and ≤10 ng/mL should undergo a prostatic biopsy or have a negative prostatic biopsy within 12 months prior to participation in the trial)
* Maximum urinary flow (Qmax) ranging between 5 to 15 mL/second with a minimum voided volume >125 mL at screening

Exclusion Criteria:

* Post void residual volume (PVR) >250 mL
* Stone in the bladder or urethra causing symptoms
* Acute or chronic prostatitis
* Interstitial cystitis / painful bladder syndrome
* Acute or recurrent urinary tract infections
* History of acute urinary retention (AUR)
* Lower urinary tract instrumentation (including prostate biopsy) within 30 days of dosing at Visit 2
* Clinical evidence of any of the following urinary tract conditions:

  1. Mullerian duct cysts
  2. Atonic, decompensated, or hypocontractile bladder
  3. Detrusor-sphincter dyssynergia (contraction of the detrusor without sphincter relaxation)
* History of any of the following pelvic conditions:

  1. Pelvic surgery or any other pelvic procedure, including radical prostatectomy, pelvic surgery for removal of malignancy, or open lower colonic or rectal surgery
  2. Pelvic radiotherapy
  3. Any prior surgical procedure of the urinary tract, including minimally invasive LUTS/BPH therapies
  4. Lower tract malignancy or trauma
* Clinically significant microscopic haematuria at screening
* History of significant renal insufficiency, defined as receiving renal dialysis or having an estimated creatinine clearance <30 mL/minute at screening
* Systolic blood pressure >180 or <90 mmHg or diastolic blood pressure >110 or <50 mmHg at screening or malignant hypertension
* Any causes other than BPH, which may affect evaluation of symptoms of urine flow (e.g. neurogenic bladder, bladder neck contracture, urethral stricture, and bladder malignancy) as judged by the Investigator
* Use of any prohibited therapies
* Elevated liver function tests at screening:

  1. Aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP) >2 times the upper limit of normal
  2. Total bilirubin >1.5 times the upper limit of normal
* QTc interval on the screening ECG >450 ms, or a family history of long QT syndrome
* Any clinically significant disorder (other than BPH) including, but not limited to, renal, haematological, gastrointestinal, endocrine, cardiac, neurological, or psychiatric disease, or any other condition, which may affect the patient's health or the outcome of the trial as judged by the Investigator
* Diagnosed cancer within the last 5 years except for adequately managed basal cell carcinoma and squamous cell carcinoma of the skin
* History of severe untreated asthma, anaphylactic reactions, or severe urticaria and/or angioedema
* Mental incapacity or language barrier precluding adequate understanding or co-operation
* History or current evidence of drug, alcohol, or substance abuse within 6 months prior to screening
* Hypersensitivity towards any component of the investigational medicinal product (IMP)
* Previous participation in any degarelix trial

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2009-08; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (47):
- United States (15):
  - Urology Centers of Alabama, PC, Homewood, Alabama
  - Coastal Clinical Research Inc, Mobile, Alabama
  - California Professional Research, Newport Beach, California
  - Genitourinary Surgical Consultants, Denver, Colorado
  - Urology Associates , PC, Englewood, Colorado
  - South Florida Medical Research, Aventura, Florida
  - Winter Park Urology Associates, Orlando, Florida
  - Pinellas Urology Inc, St. Petersburg, Florida
  - Florida Urology Partners, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Weill Cornell Medical College New York Presbyterian, New York, New York
  - Hudson Valley Urology, PC, Poughkeepsie, New York
  - Duke University Medical Center, Durham, North Carolina
  - Patient Priority Clinical Sites, LLC, Cincinnati, Ohio
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
- Belgium (2):
  - Middelheim Antwerp, Antwerp
  - UZ Brussel, Brussels
- Canada (15):
  - Can-Med Clinical Research Inc, Victoria, British Columbia
  - Dr Steinhoff Clinical Research, Victoria, British Columbia
  - Male/Female Health and Research Centre, Barrie, Ontario
  - Bramalea Medical Centre, Brampton, Ontario
  - Brandford Urology Research, Brantford, Ontario
  - Guelp Urology, Guelph, Ontario
  - Centre for Applied Urological Research, Kingston, Ontario
  - Investigational Site, North Bay, Ontario
  - Female/Male Health Centres, Oakville, Ontario
  - Mahoney Medicine Professional Corporation, Ottawa, Ontario
  - Todd Webster Ontario Inc, Owen Sound, Ontario
  - Anthony Skehan Medicine Professional Corporation, Thunder Bay, Ontario
  - The Male Health Centre, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
  - Ultra-Med Inc, Point-Claire, Quebec
- Czechia (9):
  - Urologie, Male namesti 1783, Benešov
  - Urocentrum Brno, Purkynova 35e, Brno
  - Prvni privatni chirurgicke centrum SANUS, Labská kotlina I/1220, Hradec Králové
  - Urologicka ambulance, Litomerice (Halek), Litoměřice
  - Slezska nemocnice, prospevkova organizace, Urologicke oddeleni, Opava
  - Androgeos - soukrome urologicke a andrologicke cen, Na valech 4/289, Prague
  - Urocentrum, Karlovo namesti 3, Prague
  - Urologica ambulance, Praha 10, Prague
  - Ústecké urocentrum, Ústi nad Labem (Liehne), Ústi Nad Labem
- Italy (3):
  - Urologia, A.O. San Giuseppe Moscati, Avellino, Avellino
  - Unità Operativa di Urologia, Azienda Opsedaliera Luigi Sacco, Milan
  - Unità Operativa di Urologia, Ospedale San Raffaele, Milan
- Poland (3):
  - Akademia Medyczna w Gdansku, Gdansk
  - Publiczny Specjalistyczny ZOZ, Inowrocław
  - Samodzielny Publiczny Szpital Kliniczny nr.1, Zabrze

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who met the eligibility criteria were randomised in a 1:1:1:1 manner to 1 of the 4 treatment groups in this trial. The randomisation was stratified by region (North America and Europe) and prostate volume (<30 mL and ≥30 mL). 404 patients were randomised and received a single dose of placebo, 10 mg, 20 mg, or 30 mg degarelix.
Groups:
- Placebo: Placebo: Mannitol 50 mg/mL solution. The dose was administered as a subcutaneous (s.c.) injection in the abdominal region.
- Degarelix 10 mg: Degarelix 10 mg: 10 mg degarelix, 40 mg/mL solution. The dose was administered as a s.c. injection in the abdominal region.
- Degarelix 20 mg: Degarelix 20 mg: 20 mg degarelix, 40 mg/mL solution. The dose was administered as a s.c. injection in the abdominal region.
- Degarelix 30 mg: Degarelix 30 mg: 30 mg degarelix, 40 mg/mL solution. The dose was administered as a s.c. injection in the abdominal region.
Period: Overall Study
Arm/Group | Placebo | Degarelix 10 mg | Degarelix 20 mg | Degarelix 30 mg
Started | 100 (Started: Randomised.) | 101 | 101 | 102
Full Analysis Set (FAS) | 100 (FAS: Received a dose of IMP and completed at least one post-baseline IPSS questionnaire.) | 101 | 100 (1 patient received 20 mg degarelix but had no post-baseline IPSS value and was excluded from the FAS) | 102
Actual Treatment | 98 (2 placebo patients received 30 mg degarelix) | 101 | 100 (1 patient randomised to 20 mg degarelix received 30 mg degarelix) | 105
Safety Analysis Set | 98 (Safety Analysis Set: Received a dose of Investigational Medicinal Product (IMP).) | 101 | 100 | 105
Visit 12, Month 6 | 93 (The trial was stopped when all patients had completed Visit 12, scheduled 6 months after the dosing.) | 91 | 90 | 95
Completed | 26 (End of Trial, Month 12: Patients who had completed the 12-month period when the trial was stopped.) | 24 | 22 | 20
Not Completed | 74 | 77 | 79 | 82
Not completed — Adverse Event | 0 | 1 | 4 | 4
Not completed — Withdrawal by Subject | 2 | 0 | 8 | 2
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 2 | 1 | 0
Not completed — Other/Unknown | 10 | 13 | 3 | 6
Not completed — Trial Terminated by Sponsor | 62 | 61 | 62 | 70

BASELINE CHARACTERISTICS:
Population: FAS. The efficacy analyses were based on the "as planned" treatment. Three patients deviated from the planned dosing and were included in the planned treatment groups in the FAS (i.e. not in the actual treatment groups as for the Safety Analysis Set).
Groups:
- Placebo: Placebo: Mannitol 50 mg/mL solution. The dose was administered as a s.c. injection in the abdominal region.
- Total: Total of all reporting groups
Arm/Group | Placebo | Degarelix 10 mg | Degarelix 20 mg | Degarelix 30 mg | Total
Number analyzed (Participants) | 100 | 101 | 100 | 102 | 403
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (7.86) | 64.9 (7.89) | 65.7 (7.12) | 65.4 (7.56) | 65.3 (7.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 100 | 101 | 100 | 102 | 403
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 0 | 4 | 9
  Not Hispanic or Latino | 99 | 97 | 100 | 98 | 394
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1 | 2
  Asian | 0 | 1 | 1 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 3 | 3 | 3 | 13
  White | 96 | 96 | 96 | 96 | 384
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  North America | 59 | 60 | 61 | 60 | 240
  Europe | 41 | 41 | 39 | 42 | 163
Baseline Body Mass Index (BMI) [Mean (Standard Deviation); unit: (kg/m^2)] | 28.5 (3.66) | 28.4 (3.93) | 27.9 (3.84) | 28.2 (4.81) | 28.2 (4.08)
Baseline International Prostate Symptom Scores (IPSS) [Mean (Standard Deviation); unit: units on a scale] — The IPSS questionnaire was used to assess the severity of Lower Urinary Tract Symptoms (LUTS). A detailed description of the questionnaire is provided in the Primary Outcome Measure section.
  units on a scale | 19.1 (4.38) | 19.9 (5.21) | 19.6 (4.42) | 19.8 (4.88) | 19.6 (4.73)
Baseline Total Prostate Volume (TPV) [Mean (Standard Deviation); unit: mL] — TPV was measured directly by Trans-Rectal Ultrasound (TRUS).
  mL | 41.6 (17.8) | 42.9 (18.8) | 42.3 (20.2) | 42.1 (20.2) | 42.2 (19.2)
Baseline Maximum Urinary Flow (Qmax) [Mean (Standard Deviation); unit: mL/sec] — Uroflowmetry was used according to International Continence Society (ICS) recommendation.
  mL/sec | 10.2 (2.51) | 10.3 (2.65) | 10.6 (4.58) | 10.2 (2.44) | 10.3 (3.05)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in International Prostate Symptom Score (IPSS)
Description: This outcome measure was used to assess the dose-response of the 3 degarelix dose groups in terms of severity of lower urinary tract symptoms (LUTS) and progress of the disease process, versus the placebo group. One treatment month equals 28 days.
  The IPSS questionnaire is a tool commonly used to assess the severity of LUTS, and to monitor the progress of the symptoms during treatment. It contains 7 questions regarding incomplete emptying, frequency, intermittency, urgency, weak stream, straining, and nocturia. Each question is assigned a score of 0-5 (i.e. minimum total score is 0 and the maximum score is 35), where "0" corresponds to a response of "not at all" for the first six symptoms and "none" for nocturia, and "5" corresponds to a response of "almost always" for the first six symptoms and "5 times or more" for nocturia. The IPSS also includes a question to evaluate a patient's quality of life in relation to his urinary symptoms, which is not included in the total IPSS score.
Time Frame: From Baseline to Month 3 after Dosing
Population: FAS. The "as planned" patient allocation for treatment groups was used in the efficacy analyses (please refer to the Baseline Characteristics section).
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Groups:
- Placebo: Mannitol 50 mg/mL solution. The dose was administered as a subcutaneous (s.c.) injection in the abdominal region.
- Degarelix 10 mg: Degarelix 10 mg: 10 mg degarelix, 40 mg/mL solution. The dose was administered as a subcutaneous (s.c.) injection in the abdominal region.
Arm/Group | Placebo | Degarelix 10 mg | Degarelix 20 mg | Degarelix 30 mg
Number analyzed (Participants) | 100 | 101 | 100 | 102
percentage change from baseline | -4.46 (5.34) | -5.65 (6.03) | -6.11 (5.7) | -5.88 (5.97)
Statistical Analysis 1: Comparison: Placebo vs Degarelix 30 mg; Analysis of Covariance (ANCOVA) of the change from baseline in IPSS at Month 3 in the FAS population using the Last Observation Carried Forward (LOCF) method, including the baseline IPSS as adjusting covariate and treatment group, prostate volume stratum (<30 mL and ≥30 mL), and region (North America and Europe) as factors; Test type: Superiority or Other; p = 0.0911, Step-down, Williams' extended trend test — P-value based on Williams' extended trend test of comparison vs. placebo at Month 3. No adjustment for multiple comparisons was made; Step-down procedure (starting with 30 mg vs. placebo) to identify the minimum effective dose. The step-down testing protects the type I error rate; Mean Difference (Final Values) = -1.30 — Treatment difference between "Degarelix 30 mg" and "Placebo" at Month 3
Statistical Analysis 2: Comparison: Placebo vs Degarelix 20 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0865, Step-down, Williams' extended trend test — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.44 — Treatment difference between "Degarelix 20 mg" and "Placebo" at Month 3
Statistical Analysis 3: Comparison: Placebo vs Degarelix 10 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2342, Step-down, Williams' extended trend test — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.92 — Treatment difference between "Degarelix 10 mg" and "Placebo" at Month 3

2. Secondary Outcome: Mean Change in IPSS
Description: This secondary outcome measure was used to assess the maintained dose-response of the 3 degarelix dose groups in terms of severity of LUTS and progress of the disease process, versus the placebo group.
Time Frame: From Baseline to Month 4, Month 5 and Month 6 after Dosing
Population: FAS. The "as planned" patient allocation for treatment groups was used (please refer to the Baseline Characteristics section).
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Placebo | Degarelix 10 mg | Degarelix 20 mg | Degarelix 30 mg
Number analyzed (Participants) | 100 | 101 | 100 | 102
percentage change from baseline
  Mean Percentage Change at Month 4 | -4.12 (5.65) | -5.52 (6.18) | -6.3 (6.38) | -5.64 (5.6)
  Mean Percentage Change at Month 5 | -4.34 (5.94) | -5.59 (6.89) | -6.1 (6.46) | -5.37 (5.97)
  Mean Percentage Change at Month 6 | -4.3 (5.47) | -5.42 (6.7) | -5.72 (5.59) | -5.62 (5.69)
Statistical Analysis 1: Comparison: Placebo vs Degarelix 30 mg; ANCOVA of the change from baseline in IPSS at Months 4 in the FAS population using the LOCF method, including the baseline IPSS as adjusting covariate and treatment group, prostate volume stratum (<30 mL and ≥30 mL), and region (North America and Europe) as factors; Test type: Superiority or Other; p = 0.0367, Step-down, Williams' extended trend test — P-values based on Williams' extended trend test of comparison vs. placebo at Month 4. No adjustment for multiple comparisons was made; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.62 — Treatment difference between "Degarelix 30 mg" and "Placebo" at Month 4
Statistical Analysis 2: Comparison: Placebo vs Degarelix 20 mg; ANCOVA of the change from baseline in IPSS at Month 4 in the FAS population using the LOCF method, including the baseline IPSS as adjusting covariate and treatment group, prostate volume stratum (<30 mL and ≥30 mL), and region (North America and Europe) as factors; Test type: Superiority or Other; p = 0.0231, Step-down, Williams' extended trend test — P-value based on Williams' extended trend test of comparison vs. placebo at Month 4. No adjustment for multiple comparisons was made; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.97 — Treatment difference between "Degarelix 20 mg" and "Placebo" at Month 4
Statistical Analysis 3: Comparison: Placebo vs Degarelix 10 mg; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.1638, Step-down, Williams' extended trend test — [p-value comment as in outcome 2, analysis 2]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.11 — Treatment difference between "Degarelix 10 mg" and "Placebo" at Month 4
Statistical Analysis 4: Comparison: Placebo vs Degarelix 30 mg; ANCOVA of the change from baseline in IPSS at Month 5 in the FAS population using the LOCF method, including the baseline IPSS as adjusting covariate and treatment group, prostate volume stratum (<30 mL and ≥30 mL), and region (North America and Europe) as factors; Test type: Superiority or Other; p = 0.1941, Step-down, Williams' extended trend test — P-values based on Williams' extended trend test of comparisons vs. placebo at Month 5. No adjustment for multiple comparison was made; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.14 — Treatment difference between "Degarelix 30 mg" and "Placebo" at Month 5
Statistical Analysis 5: Comparison: Placebo vs Degarelix 20 mg; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.1083, Step-down, Williams' extended trend test — P-value based on Williams' extended trend test of comparison vs. placebo at Month 5. No adjustment for multiple comparisons was made; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.54 — Treatment difference between "Degarelix 20 mg" and "Placebo" at Month 5
Statistical Analysis 6: Comparison: Placebo vs Degarelix 10 mg; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.2782, Step-down, Williams' extended trend test — [p-value comment as in outcome 2, analysis 5]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.95 — Treatment difference between "Degarelix 10 mg" and "Placebo" at Month 5
Statistical Analysis 7: Comparison: Placebo vs Degarelix 30 mg; ANCOVA of the change from baseline in IPSS at Month 6 in the FAS population using the LOCF method, including the baseline IPSS as adjusting covariate and treatment group, prostate volume stratum (<30 mL and ≥30 mL), and region (North America and Europe) as factors; Test type: Superiority or Other; p = 0.1562, Step-down, Williams' extended trend test — P-values based on Williams' extended trend test of comparison vs. placebo at Month 6. No adjustment for multiple comparisons was made; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.15 — Treatment difference between "Degarelix 30 mg" and "Placebo" at Month 6
Statistical Analysis 8: Comparison: Placebo vs Degarelix 20 mg; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; p = 0.1736, Step-down, Williams' extended trend test — P-value based on Williams' extended trend test of comparison vs. placebo at Month 6. No adjustment for multiple comparisons was made; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.24 — Treatment difference between "Degarelix 20 mg" and "Placebo" at Month 6
Statistical Analysis 9: Comparison: Placebo vs Degarelix 10 mg; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; p = 0.3132, Step-down, Williams' extended trend test — [p-value comment as in outcome 2, analysis 8]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.84 — Treatment difference between "Degarelix 10 mg" and "Placebo" at Month 6

3. Secondary Outcome: Odds Ratio (as Compared to Placebo) of Treatment Response in IPSS
Description: A 3-point reduction in IPSS score compared to baseline is defined as a clinically meaningful treatment response. Percentage of participants who met criteria for a clinically meaningful treatment response and odds ratios of treatment responses between each degarelix dose group and the placebo group are presented.
Time Frame: At Month 3, Month 4, Month 5 and Month 6 after Dosing
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Degarelix 10 mg | Degarelix 20 mg | Degarelix 30 mg
Number analyzed (Participants) | 100 | 101 | 100 | 102
percentage of participants
  3-point reduction in IPSS vs. baseline (Month 3) | 59.0 | 72.3 | 69.0 | 68.6
  3-point reduction in IPSS vs. baseline (Month 4) | 57.0 | 65.3 | 71.0 | 70.6
  3-point reduction in IPSS vs. baseline (Month 5) | 61.0 | 64.4 | 66.0 | 67.6
  3-point reduction in IPSS vs. baseline (Month 6) | 62.0 | 68.3 | 67.0 | 71.6
Statistical Analysis 1: Comparison: Placebo vs Degarelix 30 mg; Test type: Superiority or Other; p = 0.2034, Regression, Logistic — Adjustments were made for treatment group, baseline IPSS, graphical region (North America and Europe) and baseline prostate size (<30 mL and ≥30 mL). Unadjusted p-value of comparison vs. placebo at Month 3; No adjustment for multiple comparisons was made. LOCF; Odds Ratio (OR) = 1.46, 95% CI 2-sided [0.814 to 2.628] — Odds ratio of treatment response between "Degarelix 30 mg" and "Placebo" at Month 3
Statistical Analysis 2: Comparison: Placebo vs Degarelix 20 mg; Test type: Superiority or Other; p = 0.1748, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; No adjustment for multiple comparisons was made. LOCF; Odds Ratio (OR) = 1.50, 95% CI 2-sided [0.834 to 2.710] — Odds ratio of treatment response between "Degarelix 20 mg" and "Placebo" at Month 3
Statistical Analysis 3: Comparison: Placebo vs Degarelix 10 mg; Test type: Superiority or Other; p = 0.0658, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; No adjustment for multiple comparisons was made. LOCF; Odds Ratio (OR) = 1.75, 95% CI 2-sided [0.964 to 3.195] — Odds ratio of treatment response between "Degarelix 10 mg" and "Placebo" at Month 3
Statistical Analysis 4: Comparison: Placebo vs Degarelix 30 mg; Test type: Superiority or Other; p = 0.0587, Regression, Logistic — Adjustments were made for treatment group, baseline IPSS, graphical region (North America and Europe) and baseline prostate size (<30 mL and ≥30 mL). Unadjusted p-value of comparison vs. placebo at Month 4; No adjustment for multiple comparisons was made. LOCF; Odds Ratio (OR) = 1.77, 95% CI 2-sided [0.979 to 3.184] — Odds ratio of treatment response between "Degarelix 30 mg" and "Placebo" at Month 4
Statistical Analysis 5: Comparison: Placebo vs Degarelix 20 mg; Test type: Superiority or Other; p = 0.0490, Regression, Logistic — [p-value comment as in outcome 3, analysis 4]; No adjustment for multiple comparisons was made. LOCF; Odds Ratio (OR) = 1.81, 95% CI 2-sided [1.003 to 3.283] — Odds ratio of treatment response between "Degarelix 20 mg" and "Placebo" at Month 4
Statistical Analysis 6: Comparison: Placebo vs Degarelix 10 mg; Test type: Superiority or Other; p = 0.2742, Regression, Logistic — [p-value comment as in outcome 3, analysis 4]; No adjustment for multiple comparisons was made. LOCF; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.774 to 2.464] — Odds ratio of treatment response between "Degarelix 10 mg" and "Placebo" at Month 4
Statistical Analysis 7: Comparison: Placebo vs Degarelix 30 mg; Test type: Superiority or Other; p = 0.4206, Regression, Logistic — Adjustments were made for treatment group, baseline IPSS, graphical region (North America and Europe) and baseline prostate size (<30 mL and ≥30 mL). Unadjusted p-value of comparison vs. placebo at Month 5; No adjustment for multiple comparisons was made. LOCF; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.706 to 2.304] — Odds ratio of treatment response between "Degarelix 30 mg" and "Placebo" at Month 5
Statistical Analysis 8: Comparison: Placebo vs Degarelix 20 mg; Test type: Superiority or Other; p = 0.5494, Regression, Logistic — [p-value comment as in outcome 3, analysis 7]; No adjustment for multiple comparisons was made. LOCF; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.664 to 2.160] — Odds ratio of treatment response between "Degarelix 20 mg" and "Placebo" at Month 5
Statistical Analysis 9: Comparison: Placebo vs Degarelix 10 mg; Test type: Superiority or Other; p = 0.7586, Regression, Logistic — [p-value comment as in outcome 3, analysis 7]; No adjustment for multiple comparisons was made. LOCF; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.609 to 1.975] — Odds ratio of treatment response between "Degarelix 10 mg" and "Placebo" at Month 5
Statistical Analysis 10: Comparison: Placebo vs Degarelix 30 mg; Test type: Superiority or Other; p = 0.1946, Regression, Logistic — Adjustments were made for treatment group, baseline IPSS, graphical region (North America and Europe) and baseline prostate size (<30 mL and ≥30 mL). Unadjusted p-value of comparison vs. placebo at Month 6; No adjustment for multiple comparisons was made. LOCF; Odds Ratio (OR) = 1.49, 95% CI 2-sided [0.816 to 2.717] — Odds ratio of treatment response between "Degarelix 30 mg" and "Placebo" at Month 6
Statistical Analysis 11: Comparison: Placebo vs Degarelix 20 mg; Test type: Superiority or Other; p = 0.5380, Regression, Logistic — [p-value comment as in outcome 3, analysis 10]; No adjustment for multiple comparisons was made. LOCF; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.667 to 2.174] — Odds ratio of treatment response between "Degarelix 20 mg" and "Placebo" at Month 6
Statistical Analysis 12: Comparison: Placebo vs Degarelix 10 mg; Test type: Superiority or Other; p = 0.4263, Regression, Logistic — [p-value comment as in outcome 3, analysis 10]; No adjustment for multiple comparisons was made. LOCF; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.702 to 2.308] — Odds ratio of treatment response between "Degarelix 10 mg" and "Placebo" at Month 6

4. Secondary Outcome: Mean Percentage Change in Total Prostate Volume (TPV)
Description: TPV was measured directly by standardised trans-rectal ultrasound (TRUS).
Time Frame: From Baseline to Month 3 and Month 6 after Dosing
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Placebo | Degarelix 10 mg | Degarelix 20 mg | Degarelix 30 mg
Number analyzed (Participants) | 100 | 101 | 100 | 102
percentage change from baseline
  Mean Percentage Change at Month 3 | 3.15 (23.3) | -1.46 (32.7) | -0.252 (24.5) | 0.188 (24.4)
  Mean Percentage Change at Month 6 | 3.96 (29.3) | 1.57 (31) | 2.35 (26.5) | -0.0112 (20.9)
Statistical Analysis 1: Comparison: Placebo vs Degarelix 30 mg; Test type: Superiority or Other; p = 0.4607, ANCOVA — No adjustment for multiple comparisons was made. Unadjusted p-value of comparison vs. placebo at Month 3; ANCOVA with baseline TPV as covariate and treatment group, region (North America,Europe) and prostate volume stratum (<30 mL,≥30 mL) as factors. LOCF; Mean Difference (Final Values) = -2.76, 95% CI 2-sided [-10.113 to 4.590] — Treatment difference between "Degarelix 30 mg" and "Placebo" at Month 3
Statistical Analysis 2: Comparison: Placebo vs Degarelix 20 mg; Test type: Superiority or Other; p = 0.3876, ANCOVA — No adjustment for multiple comparisons was made. Unadjusted p-value of comparison vs. placebo at Month 3; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -3.24, 95% CI 2-sided [-10.614 to 4.128] — Treatment difference between "Degarelix 20 mg" and "Placebo" at Month 3
Statistical Analysis 3: Comparison: Placebo vs Degarelix 10 mg; Test type: Superiority or Other; p = 0.2548, ANCOVA — No adjustment for multiple comparisons was made. Unadjusted p-value of comparison vs. placebo at Month 3; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -4.28, 95% CI 2-sided [-11.650 to 3.096] — Treatment difference between "Degarelix 10 mg" and "Placebo" at Month 3
Statistical Analysis 4: Comparison: Placebo vs Degarelix 30 mg; Test type: Superiority or Other; p = 0.5652, ANCOVA — No adjustment for multiple comparisons was made. Unadjusted p-value of comparison vs. placebo at Month 6; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -2.20, 95% CI 2-sided [-9.729 to 5.322] — Treatment difference between "Degarelix 30 mg" and "Placebo" at Month 6
Statistical Analysis 5: Comparison: Placebo vs Degarelix 20 mg; Test type: Superiority or Other; p = 0.7502, ANCOVA — No adjustment for multiple comparisons was made. Unadjusted p-value of comparison vs. placebo at Month 6; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -1.22, 95% CI 2-sided [-8.768 to 6.322] — Treatment difference between "Degarelix 20 mg" and "Placebo" at Month 6
Statistical Analysis 6: Comparison: Placebo vs Degarelix 10 mg; Test type: Superiority or Other; p = 0.6089, ANCOVA — No adjustment for multiple comparisons was made. Unadjusted p-value of comparison vs. placebo at Month 6; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -1.97, 95% CI 2-sided [-9.513 to 5.581] — Treatment difference between "Degarelix 10 mg" and "Placebo" at Month 6

5. Secondary Outcome: Mean Change in Maximum Urinary Flow (Qmax)
Description: Urinary flow rate (mL/second) was measured using uroflowmetry performed according to the recommendation from the International Continence Society (ICS).
Time Frame: From Baseline to Month 3 and Month 6 after Dosing
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Placebo | Degarelix 10 mg | Degarelix 20 mg | Degarelix 30 mg
Number analyzed (Participants) | 100 | 101 | 100 | 102
percentage change from baseline
  Mean Percentage Change at Month 3 | 0.652 (3.8) | 0.564 (5.08) | 0.626 (5.68) | 0.723 (3.91)
  Mean Percentage Change at Month 6 | 1.04 (5.34) | 0.516 (4.85) | 0.582 (5.43) | 1.43 (5.29)
Statistical Analysis 1: Comparison: Placebo vs Degarelix 30 mg; Test type: Superiority or Other; p = 0.8511, ANCOVA — No adjustment for multiple comparisons was made. Unadjusted p-value of comparison vs. placebo at Month 3; ANCOVA with baseline Qmax as covariate and treatment group, region (North America,Europe) and prostate volume stratum (<30 mL,≥30 mL) as factors.LOCF; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-1.068 to 1.294] — Treatment difference between "Degarelix 30 mg" and "Placebo" at Month 3
Statistical Analysis 2: Comparison: Placebo vs Degarelix 20 mg; Test type: Superiority or Other; p = 0.6331, ANCOVA — No adjustment for multiple comparisons was made. Unadjusted p-value of comparison vs. placebo at Month 3; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = 0.29, 95% CI 2-sided [-0.900 to 1.477] — Treatment difference between "Degarelix 20 mg" and "Placebo" at Month 3
Statistical Analysis 3: Comparison: Placebo vs Degarelix 10 mg; Test type: Superiority or Other; p = 0.9090, ANCOVA — No adjustment for multiple comparisons was made. Unadjusted p-value of comparison vs. placebo at Month 3; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-1.113 to 1.250] — Treatment difference between "Degarelix 10 mg" and "Placebo" at Month 3
Statistical Analysis 4: Comparison: Placebo vs Degarelix 30 mg; Test type: Superiority or Other; p = 0.5469, ANCOVA — No adjustment for multiple comparisons was made. Unadjusted p-value of comparison vs. placebo at Month 6; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = 0.42, 95% CI 2-sided [-0.956 to 1.802] — Treatment difference between "Degarelix 30 mg" and "Placebo" at Month 6
Statistical Analysis 5: Comparison: Placebo vs Degarelix 20 mg; Test type: Superiority or Other; p = 0.7906, ANCOVA — No adjustment for multiple comparisons was made. Unadjusted p-value of comparison vs. placebo at Month 6; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-1.576 to 1.200] — Treatment difference between "Degarelix 20 mg" and "Placebo" at Month 6
Statistical Analysis 6: Comparison: Placebo vs Degarelix 10 mg; Test type: Superiority or Other; p = 0.5757, ANCOVA — No adjustment for multiple comparisons was made. Unadjusted p-value of comparison vs. placebo at Month 6; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-1.773 to 0.987] — Treatment difference between "Degarelix 10 mg" and "Placebo" at Month 6

ADVERSE EVENTS:
Time Frame: This was a single dose trial and adverse events were recorded from signed informed consent up to a maximum of 12 months after the dose. However, the trial was stopped when all patients had completed the visit scheduled 6 months after the dosing.
Description: Adverse events were evaluated at each visit. The safety analyses were based on the actual treatment. Three patients did not receive their randomised treatment: 2 patients randomised to placebo received 30 mg, and 1 patient randomised to 20 mg received 30 mg degarelix. They were included in the actual treatment group in the safety analysis set.
Arm/Group | Placebo | Degarelix 10 mg | Degarelix 20 mg | Degarelix 30 mg
Serious Adverse Events (participants affected / at risk) | 2/98 | 8/101 | 2/100 | 7/105
Other Adverse Events (participants affected / at risk) | 31/98 | 35/101 | 39/100 | 56/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=98) | Degarelix 10 mg (N=101) | Degarelix 20 mg (N=100) | Degarelix 30 mg (N=105)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess intestinal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coagulation time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Adenosquamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carotid sinus syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=98) | Degarelix 10 mg (N=101) | Degarelix 20 mg (N=100) | Degarelix 30 mg (N=105)
Injection site erythema (General disorders) | 0 (0) | 11 (11) | 14 (14) | 18 (18)
Injection site pain (General disorders) | 0 (0) | 2 (2) | 10 (10) | 18 (19)
Injection site induration (General disorders) | 0 (0) | 6 (6) | 7 (7) | 11 (11)
Hypertension (Vascular disorders) | 7 (8) | 6 (6) | 4 (5) | 9 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 5 (5) | 5 (5) | 5 (6)
Prostatic specific antigen increased (Investigations) | 6 (6) | 4 (4) | 5 (6) | 6 (6)
Nasopharyngitis (Infections and infestations) | 5 (5) | 7 (8) | 2 (2) | 5 (5)
Hot flush (Vascular disorders) | 1 (2) | 1 (1) | 4 (4) | 8 (10)
Influenza (Infections and infestations) | 5 (5) | 5 (5) | 3 (3) | 5 (5)
Headache (Nervous system disorders) | 5 (5) | 3 (3) | 3 (3) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
Following the planned 6-month interim analysis when all patients had completed the visit scheduled 6 months after dosing, a decision was taken to stop the trial since the primary efficacy endpoint was not met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.